CLINICAL TRIAL: NCT04127279
Title: Stress Relief Properties of a Cosmetic Routine: Psychobiological Evidence
Brief Title: Stress Relief Properties of a Cosmetic Routine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Parma (Other)
Responsible Party: Principal Investigator, Elena Giovanna Bignami, full professor, University of Parma
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 46700 18122017
Record Dates: First submitted 2019-09-26; First posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Stress Physiology; Stress, Psychological
Keywords: autonomic nervous system; HPA axis; anxiety; non verbal behavior
MeSH Terms: conditions — Stress, Psychological; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enriched Cream (Experimental): The enriched cream is self-administered and contains a blend of 4 essential oils, namely Juniperus phoenicea gum extract, Copaifera officinalis resin, Aniba rosaeodora wood oil and Juniperus virginiana oil.
  Interventions: Biological: Cream
- Placebo Cream (Active Comparator): Cream devoid of essential oils, self-administered
  Interventions: Biological: Cream

INTERVENTIONS:
Biological: Cream — The enriched cream is self-administered and contains a blend of 4 essential oils, namely Juniperus phoenicea gum extract, Copaifera officinalis resin, Aniba rosaeodora wood oil and Juniperus virginiana oil.
  The placebo cream is devoid of the essential oils

SUMMARY:
Everyday life psychosocial challenges may negatively impact health and well-being, contributing to the onset and/or progression of psychological and psychosomatic disorders. Pharmacological treatments can moderate our stress response, but they usually bring about addiction/tolerance and a number of other side effects. Therefore, it is relevant to identify alternative stress relief strategies that are devoid of these unwanted drawbacks. Moreover, the effects of such alternative interventions should be objectively quantified by means of reliable psychobiological parameters. The goal of this study was to quantify the acute and persistent effects of a cosmetic routine based on the self-administration of a cream enriched with essential oils, namely Juniperus Phoenicea gum extract, Copaifera Officinalis resin, Aniba Rosodora wood oil, and Juniperus Virginiana. This aim was achieved by measuring the (re-)activity of the autonomic nervous system (via heart variability indexes) and the hypothalamic-pituitary-adrenocortical axis (via salivary cortisol levels), as well as through psychometric and behavioral assessments.

Participants' informed consent signature for adhesion at the study was initially requested. With their acceptance, parameters were recorded anonimously, identified by their initials and an alphanumeric code.

Data were transferred on Excel worksheets, utilized for descriptive analysis related at every variable. All statistical analyses were performed using SPSS 25 software package and statistical significance was set at p<0.05.

DETAILED DESCRIPTION:
Everyday life psychosocial challenges may negatively impact health and well-being, contributing to the onset and/or progression of psychological and psychosomatic disorders. Pharmacological treatments can moderate our stress response, but they usually bring about addiction/tolerance and a number of other side effects. Therefore, it is relevant to identify alternative stress relief strategies that are devoid of these unwanted drawbacks. Moreover, the effects of such alternative interventions should be objectively quantified by means of reliable psychobiological parameters.

The goal of this study was to quantify the acute and persistent effects of a cosmetic routine based on the self-administration of a cream (DAVC) enriched with essential oils, namely Juniperus Phoenicea gum extract, Copaifera Officinalis resin, Aniba Rosodora wood oil, Juniperus Virginiana. This aim was achieved by measuring the (re-)activity of the autonomic nervous system (via heart variability indexes) and the hypothalamic-pituitary-adrenocortical axis (via salivary cortisol levels), as well as through psychometric and behavioral assessments.

Fourty women, 25-50 years old, were instructed for a correct mode of self administration of the cream. On day 0, women came to the lab and were instrumented for electrocardiographic signal (ECG) recordings. Initially, a 10-min ECG was collected in resting conditions (baseline). Then, two 20-min ECGs were recorded, each following the self-administration (3-min duration) of the DAVC and a placebo cream (PLAC), in a randomized order. At the end of the baseline and the two post-cream administration recordings, saliva samples were collected. From day 1 to 28, subjects self-administered (at home, twice a day, at wake-up and bed time) either DAVC (n=20) or PLAC (n=20).

On day 29, they returned to the lab and ECGs and underwent a stress test (Trier Social Stress Test, TSST). The test lasted 10 min and consisted in a stress interview (5 min), immediately followed by an arithmetic task. ECGs were collected in baseline (10 min), test (10 min), and recovery (20 min) phases. Saliva samples were collected at the end of the baseline and the middle and the end of the recovery phase. The subjects filled a number of psychological questionnaires, including Profile of Mood States (POMS, on day 0 and 29) and STAI-Y1 (on day 29). In addition, subjects were videorecorded during the TSST, in order to quantify their non verbal behavior patterns (via ECSI).

A single, self-administration of DAVC (day 0) produced a significant, acute potentiation of parasympathetic neural modulation (HF index: 25% increase as to baseline), whereas PLAC produced only a modest change (3% increase). DAVC provoked a modest (10%), non significant reduction of cortisol levels, which was similar to that induced by PLAC.

Prolonged DAVC self-administration (4 weeks) produced: (i) a significant inhibition of stress-induced cortisol elevation on day 29 (55% increase as compared to pre-stress value in DAVC group, 75% in PLAC group); (ii) a significant improvement of mood profile (POMS test) on day 29 compared to day 0; (iii) a reduction of perceived anxiety (STAI-Y1 score) at the end of the TSST; (iv) significantly lower scores of behavioral patterns linked to anxiety, motivational conflict and avoidance and higher scores of affiliation during the TSST, as compared to PLAC group.

These autonomic neural, neuroendocrine and psychological data suggest that a cream enriched with essential oils has both acute and long-term stress-reduction effects on human psychophysiology. Acute effects involve a potentiation of the parasympathetic component of autonomic neural regulation, which is usually associated with well-being, relaxation and resilience. The long-term effects point to a generalized stress-relief property, involving both the hormonal and psychological sides of stress adaptation.

ELIGIBILITY:
Inclusion Criteria:

* female gender
* 25 to 50 years old

Exclusion Criteria:

* current or past neurological, psychiatric, and cardiac disorders
* cognitive impairment
* substance or alcohol abuse or dependence
* recent (last 12 months) traumatic events such as a death in the family, serious accident, job firing or divorce
* caregiving (last 12 months) a family member with serious pathology or disability
* current psychotropic or contraceptive drug use

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
Acute autonomic stress responsivity (heart rate, HR) to cream self-administration | ECG recorded just before (for 10 minutes) the self-administration of the enriched and placebo creams (day 0)
  Mean HR, measured as bpm (beats per minute)
Acute autonomic stress responsivity (heart rate, HR) to cream self-administration | ECG recorded just after (for 20 minutes) the self-administration of the enriched and placebo creams (day 0)
  Mean HR, measured as bpm (beats per minute)
Acute autonomic stress responsivity (HF, vagal input to the heart) to cream self-administration | ECG recorded just before (for 10 minutes) the self-administration of the enriched and placebo creams (day 0)
  High frequency component power (HF) of the RR interval spectrum (n.u.)
Acute autonomic stress responsivity (HF, vagal input to the heart) to cream self-administration | ECG recorded just after (for 20 minutes) the self-administration of the enriched and placebo creams (day 0)
  High frequency component power (HF) of the RR interval spectrum (n.u.)
Acute HPA axis stress responsivity to cream self-administration | Samples obtained just before the self-administration of the enriched and placebo creams
  Determined by means of salivary cortisol levels (pg/ml)
Acute HPA axis stress responsivity to cream self-administration | Samples obtained after (20 min) the self-administration of the enriched and placebo creams
  Determined by means of salivary cortisol levels (pg/ml)
Acute HPA axis stress responsivity to the psychosocial stress test | Samples obtained just before the psychosocial stress test
  Determined by means of salivary cortisol levels
Acute HPA axis stress responsivity to the psychosocial stress test | Samples obtained after (10 minutes) the psychosocial stress test
  Determined by means of salivary cortisol levels
Acute HPA axis stress responsivity to the psychosocial stress test | Samples obtained after (30 minutes) the psychosocial stress test
  Determined by means of salivary cortisol levels

SECONDARY OUTCOMES:
Perceived stress | Before (day -2) the 4-week time period (day 0 to 28) during which subjects self-administered twice daily (at wake up time and bed time) the cream
  Determined via the Perceived Stress Scale (PSS) questionnaire. It is a measure of the degree to which situations in one's life are appraised as stressful. Items are designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives. The 10 questions that compose this test are related to feelings and thoughts experienced during the last month. In each case, respondents are asked how often they felt a certain way.
  For each question, they had to choose from the following alternatives:
  0=never, 1=almost never, 2=sometimes, 3=fairly often, 4=very often.
  The PSS score was determined by following these directions:
  First, the scores for questions 4, 5, 7, and 8 were reversed.
  On these 4 questions, the scores were changed like this:
  0 = 4, 1 = 3, 2 = 2, 3 = 1, 4 = 0.
  Then scores were added up for each item to get a total. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Perceived stress | After (day 29) the 4-week time period (day 0 to 28) during which subjects self-administered twice daily (at wake up time and bed time) the cream
  Determined via the Perceived Stress Scale (PSS) questionnaire. It is a measure of the degree to which situations in one's life are appraised as stressful. Items are designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives. The 10 questions that compose this test are related to feelings and thoughts experienced during the last month. In each case, respondents are asked how often they felt a certain way.
  For each question, they had to choose from the following alternatives:
  0=never, 1=almost never, 2=sometimes, 3=fairly often, 4=very often.
  The PSS score was determined by following these directions:
  First, the scores for questions 4, 5, 7, and 8 were reversed.
  On these 4 questions, the scores were changed like this:
  0 = 4, 1 = 3, 2 = 2, 3 = 1, 4 = 0.
  Then scores were added up for each item to get a total. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Profile of mood states | Before (day -2) the 4-week time period (day 0 to 28) during which subjects self-administered twice daily (at wake up time and bed time) the cream
  Determined via the Profile of Mood States (POMS) questionnaire. It is a rating scale that measures 6 distinct mood states, namely tension-anxiety (TA), depression-dejection (DD), anger-hostility (AH), fatigue-inertia (FI), confusion-bewilderment (CB), and vigor-activity (VA). Subjects are asked to report the intensity of these six different dimensions of mood as they felt them during the last week. Subjects self report on each of these areas using a 5-point Likert scale (0=not at all, 1=a little, 2=moderately, 3=quite a lot, 4=extremely). An overall score of mood profile (POMS score) can be drawn by summing the scores obtained in each of the five "negative" factors and subtracting the single positive factor (VA).
Profile of mood states | After (day 29) the 4-week time period (day 0 to 28) during which subjects self-administered twice daily (at wake up time and bed time) the cream
  Determined via the Profile of Mood States (POMS) questionnaire. It is a rating scale that measures 6 distinct mood states, namely tension-anxiety (TA), depression-dejection (DD), anger-hostility (AH), fatigue-inertia (FI), confusion-bewilderment (CB), and vigor-activity (VA). Subjects are asked to report the intensity of these six different dimensions of mood as they felt them during the last week. Subjects self report on each of these areas using a 5-point Likert scale (0=not at all, 1=a little, 2=moderately, 3=quite a lot, 4=extremely). An overall score of mood profile (POMS score) can be drawn by summing the scores obtained in each of the five "negative" factors and subtracting the single positive factor (VA).
Behavioral coping style | During the psychosocial stress test (PST, day 29)
  Determined via the quantification of 37 different patterns of non-verbal behavior. The recording session (10-min psychosocial stress) was divided into successive 15-second sample intervals. The instant of time at the end of each sample interval, referred to as the "sample point", was identified by a beeper. On the instant of each sample point, the observer recorded whether or not the behavior pattern had occurred during the preceding sample interval. The score of each behavior for each subject was expressed as the proportion of all sample intervals during which that behavior occurred.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Sgoifo, PhD, Principal Investigator — University of Parma; Luca Carnevali, PhD, Principal Investigator — University of Parma
Locations (1):
- University of Parma, Parma, Italy